CLINICAL TRIAL: NCT05160181
Title: Impact of Yogotherapeutics in Consultation on Chronic Pains' Patients
Brief Title: Impact of Yogotherapeutics on Chronic Pains' Patients
Acronym: YOGADO
Status: Completed | Type: Observational
Sponsor: Hôpital NOVO (Other)
Responsible Party: Sponsor
Other Study IDs: CHRD1119
Record Dates: First submitted 2021-12-03; First posted 2021-12-16 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2022-04

CONDITIONS: Chronic Pain
Keywords: Chronic Pain; Yogatherapeutics
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Yogatherapy: Retrospective study on medical file of patients seen in consultation for chronic pain with prescription of Yogatherapy
  Interventions: Other: Yogatherapy

INTERVENTIONS:
Other: Yogatherapy — Description: Retrospective study on medical file of patients seen in consultation for chronic pain with prescription of Yogatherapy

SUMMARY:
In a context where yoga is more and more popularized in France and in Europe, and where Yogatherapy (as complementary medicine) begins to make its place in the care of patients in French hospitals, it seems interesting to study the impact of yoga in the chronic pain patient treated in a specific pain consultation by this non-pharmacological approach, and accessible.

DETAILED DESCRIPTION:
Yoga is a discipline that has its origins in India for nearly 5,000 years, and which aims to bring physical, mental and spiritual well-being through postures, stretching, breathing exercises and meditation.

Non-invasive and having very few side effects, this approach allows the practitioner to reclaim their body, to know themselves better, to accept their limits, to respect them and to empower themselves in their care and pathology.

More and more studies are now looking at the positive effect of yoga whether it is on stress by demonstrating the drop in cortisol in participants, or on the reduction of symptoms of depression, improvement of immune function, or pain.

To our knowledge, no study of the impact of yoga for analgesic treatment has been carried out in France.

Through this retrospective study, the investigators wish to demonstrate a reduction in pain and / or an improvement in the quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Patient ≥ 18 years old,
* Seen in consultation for chronic pain with implementation of Yogatherapy,

Exclusion Criteria:

* Patient < 18 years old,
* No indication for Yogatherapy treatment (Severe cognitive disorder / Major unbalanced psychological disorder),
* Trauma pathology and / or acute fracture in progress,
* Patient refusal to participate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients seen in consultation for chronic pain and with prescription of Yogatherapy
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2021-09-13 (Actual); Primary Completion 2022-06-28 (Actual); Study Completion 2022-06-28 (Actual)

PRIMARY OUTCOMES:
Evolution of the patient's pain | Between the 1st and the 5th consultation, an average of 3 to 5 month
  The evolution of the patient's pain is assessed by comparing the pain between the 1st and the 5th consultation, using a numerical scale from 0 to 10 points (0 = no pain and 10 = maximum pain imaginable)

SECONDARY OUTCOMES:
Evolution of the patient's pain over time | Between the 1st and the 5th consultation, an average of 3 to 5 month
  The evolution of the patient's pain is assessed by comparing the pain between the 1st and the last consultation (number 10 maximum), using a numerical scale from 0 to 10 points (0 = no pain and 10 = maximum pain imaginable)
Improvement of patient's sleep | Between the 1st and the last consultation, an average of 5 to 10 month
  The impact of pain on sleep is evaluated by questioning the patient at the first and last consultation (number 10 maximum) The answer to the question is YES or NO
Evolution of the patient's quality of life | Between the 1st and the last consultation, an average of 5 to 10 month
  The quality of life is assessed at all visits, by questioning patient, on the following elements: work, daily activities, mood…. to obtain a score on a numerical scale between 0 and 10
  Results are interpreted as following : EN ≤ 5 = Very degraded, 6 ≥ EN ≤ 7 = Degraded and EN > 7 = Normal)
Evolution of the patient's therapeutic | Between the 1st and the last consultation, an average of 5 to 10 month
  The evolution of the therapeutic is evaluated by questioning the patient at the first and last consultation (number 10 maximum) about their treatment: treatment name, indication, dosage, number of doses per day, decrease or increase for each treatment ……. to see if there is a decrease or not in the patient's therapies.

CONTACTS AND LOCATIONS:
Overall Officials: Jocelyne BOREL-KUHNER, Principal Investigator — Hospital René Dubos,
Locations (1):
- Departement of Chronic Pain Consultation, Hospital René Dubos,, Pontoise, France